CLINICAL TRIAL: NCT00398957
Title: An Open Label Evaluation of the Dose Proportionality of Dilaudid SR (OROS� Hydromorphone HCL) Tablets 8mg, 16mg, 32mg, and 64mg
Brief Title: An Open-Label Evaluation of the Dose Proportionality of OROS� Hydromorphone HCL Tablets 8mg, 16mg, 32mg, 64mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR011611
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Analgesia
Keywords: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Naltrexone

INTERVENTIONS:
Drug: OROS® Hydromorphone HCL; OROS® Dilaudid; Dilaudid SR (slow release); Naltrexone (an opioid antagonist).

SUMMARY:
The primary objective of this study was to examine the OROSÂ® Hydromorphone HCL pharmacokinetic (the way a drug enters and leaves the blood and tissues over time) profile for dose proportionality after administration of 8mg, 16mg, 32mg and 64 mg tablets.

DETAILED DESCRIPTION:
This was a randomized (patients are assigned different treatments based on chance), open-label, four-way crossover study performed in normal, healthy adult patients. Each patient received the following orally administered treatments of OROS® Hydromorphone HCL (a different treatment during each dosing phase): Treatment A: 8mg; Treatment B: 16mg; Treatment C: 32mg; Treatment D: 64mg; A naltrexone 50mg dose was administered 12 hours prior to, at the time of, and 12 after study drug administration; Patients received a fourth dose of naltrexone 50mg 24 hours after the 64mg study drug administration. There was a 7-day washout period between study drug dosing phases.Venous blood sampling times were 0 (prior to dosing), 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, and 48 hours after each study drug administration. Three additional blood samples (at 56, 64, and 72 hours after dosing of study drug) were drawn from those patients receiving the 64 mg tablets; LC/MS/MS (Liquid Chromatography/Mass Spectroscopy/Mass Spectroscopy) techniques were employed for the analysis of plasma hydromorphone concentrations.The primary endpoints of interest were: Area under the concentration-time curve from zero to infinity; Area under the concentration-time curve from zero to time t; Peak plasma concentration; the secondary endpoint parameters were: Time to peak plasma concentration; Terminal half-life. OROS hydromorphone HCL tablets of 8mg, 16mg, 32mg, and 64mg were given orally, a different dosing treatment during each dosing phase. One naltrexone HCL 50mg tablet was given orally 12 hours prior to, at the time of, and 12 hours after hydromorphone administration during each dosing phase. Patient received a fourth dose of naltrexone 50mg 24 hours following the 64mg study drug administration; It was a four week treatment and there was a seven-day washout period between dosing phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients were non-smoking, healthy volunteers with body weight between 135 and 220 pounds and within +/- 10% of their recommended weight range for their height and body frame according to the Metropolitan Height and Weight Tables
* Patients had a negative baseline urine screen for drugs of abuse
* Patients did not have any clinically significant deviations from normal in any laboratory test value.

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone or naltrexone
* Patient with any gastrointestinal disorder that may affect the absorption of orally administered drugs
* Patients with depressed respiratory function
* Patient with impaired renal or hepatic function
* Patient with dependence to opiates
* pregnant or breast feeding
* Female patients of child bearing potential must have a negative pregnancy test each week prior to administration of study drug and required to be following a medically rhydromorphoneadministrationnaltrexone recognized contraceptive program prior to and during the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoints for the statistical evaluations of the study drug were: Area Under the Concentration-Time Curve from 0 to Infinity, Area Under the Concentration-Time Curve from 0 to time t and Peak Plasma Concentration.

SECONDARY OUTCOMES:
The secondary endpoints were the pharmacokinetic parameters for the study drug: Time to Peak Plasma Concentration and Terminal half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Derived] Sathyan G, Xu E, Thipphawong J, Gupta SK. Pharmacokinetic investigation of dose proportionality with a 24-hour controlled-release formulation of hydromorphone. BMC Clin Pharmacol. 2007 Feb 2;7:3. doi: 10.1186/1472-6904-7-3. PMID 17270058